CLINICAL TRIAL: NCT00689260
Title: A Randomized, Multicenter, 3 Month Phase IV Study to Evaluate the Effect on Subject Adherence With Injection Schedule by Using the Easypod™ rhGH Delivery Device
Brief Title: Easypod United States User Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 28358
Record Dates: First submitted 2008-05-22; First posted 2008-06-03 (Estimated); Results first posted 2010-07-20 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Log Aware (Active Comparator): Dose Log Aware (patient is aware that the device records their injection information) Half the subjects in the log aware arm will complete a diary. The other half in the log aware arm will not complete the diary.
  Interventions: Device: easypod
- 2 - Log Unaware (Active Comparator): Dose Log Unaware (patient is not aware that the device records their injection information) Half the subjects in the log unaware arm will complete a diary. The other half in the log unaware arm will not complete the diary.
  Interventions: Device: easypod

INTERVENTIONS:
Device: easypod — Subjects is aware that the device records injection information that can be viewed by user
  Arms: 1 - Log Aware
Device: easypod — Subjects is not aware that the device records injection information that can be viewed by user
  Arms: 2 - Log Unaware

SUMMARY:
This study will help to determine whether an injection log on a recombinant human growth hormone (rhGH) delivery device improves subjects' adherence with injection schedules. Adherence will be compared between a group of subjects who are aware of the injection log on the easypod™ rhGH delivery device and a group of subjects who are not aware of the easypod™ injection log. It is the study hypothesis that subject non-adherence rate is different for those who are aware of the injection log capability versus those who are unaware of the injection log capability. Subject perception will also be evaluated by comparing the ease and convenience of use and subject preference for the easypod™ compared to two other rhGH pen injection devices.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female from 10 to 18 years of age, inclusive, with open epiphyses
* Have GH deficiency diagnosed by treating pediatric endocrinologist for at least 6 months
* Be undergoing rhGH treatment via self-injection using the Lilly Humatrope® or Pfizer Genotropin® pen injection device for at least 6 months
* Be willing and able to comply with the protocol for the duration of the trial
* Have access to the Internet
* Be able to read, speak and understand English
* If female of childbearing potential, have a negative urine pregnancy test at Screening and use an acceptable form of birth control during the trial, including abstinence, a hormonal contraceptive, intrauterine device, diaphragm with spermicide, or condom with spermicide

Exclusion Criteria:

* Known allergy or hypersensitivity to rhGH or prescribed diluent (0.3% metacresol for click.easy® cartridge)
* Severe illness during the previous 6 months
* Active malignancy (except non-melanomatous skin malignancies)
* Diabetes mellitus (type I or II)
* Pregnancy or lactation
* Any medical condition that, in the opinion of the Investigator, would jeopardize the subject's safety following exposure to the investigational device
* Participation in any other investigational study during the duration of participation in this trial

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, MD, Study Director — EMD Serono, Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- US Medical Information, Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 Subjects were randomized from 14 Clinics in the US from March 2008 through January 2009. One subject withdrew consent prior to first dose. Recruitment was ended early due to slow enrollment.
Pre-assignment Details: Screening and randomization took place at Visit 1 (Study Day 1) which consisted of informed consent, medical/disease history, physical exam and laboratory assessments.
Groups:
- Log Aware: Dose Log Aware and Daily Diary Enabled
- Log Unaware: Dose Log UnaAware and Daily Diary Disabled
Period: Overall Study
Arm/Group | Log Aware | Log Unaware
Started | 21 | 21
Completed | 19 | 21
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Log Aware | Log Unaware | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 21 | 42
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (1.50) | 13.0 (2.56) | 12.7 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percent rhGH Injections Missed During the Treatment Period (Based on the Easypod™ Injection Log)
Time Frame: 90 Days
Population: The modified full analysis set includes all randomized subjects who received at least one injection using the easypod device and had valid device data. Seven subjects who had damaged devices or incorrect device setting were excluded from this analysis set.
Measure: Median (Full Range); unit: Percent of injections missed
Arm/Group | Log Aware | Log Unaware | Total
Number analyzed (Participants) | 15 | 20 | 35
Percent of injections missed | 20 [0 to 71.7] | 19.46 [1.1 to 90.9] | 20 [0 to 90.9]
Statistical Analysis 1: Comparison: Log Aware vs Log Unaware; P-Value based on two-sided Wilcoxon rank-sum test for difference in medians between log aware and log unaware; Test type: Superiority or Other; p = 0.908, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Subjects Perception of Easypod Ease of Use Compared to Two Other rhGH Pen Injection Devices
Time Frame: 90 Days
Population: The modified full analysis set includes all randomized subjects who received at least one injection using the Easypod device and had valid device data. In addition, this total of 35 subjects was divided into 2 groups, Humatrope and Genotropin, based on their previous rhGH use.
Measure: Number; unit: Participants
Groups:
- Humatrope: Subjects previously using the Lilly Humatrope
- Genotropin: Subjects previously using the Pfizer Genotropin
Arm/Group | Humatrope | Genotropin | Total
Number analyzed (Participants) | 16 | 19 | 35
Participants
  Strongly Agree | 5 | 5 | 10
  Agree | 1 | 3 | 4
  Neutral | 0 | 4 | 4
  Disagree | 3 | 1 | 4
  Strongly Disagree | 2 | 3 | 5
  Missing | 5 | 3 | 8

3. Secondary Outcome: Subject Perceptions of Easypod: Storage Convenience Compared to Two Other rhGH Pen Injection Devices.
Time Frame: 90 Days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Humatrope | Genotropin | Total
Number analyzed (Participants) | 16 | 19 | 35
Participants
  Very Convenient | 3 | 7 | 10
  Convenient | 3 | 5 | 8
  Neutral | 5 | 3 | 8
  Not Very Convenient | 0 | 0 | 0
  Not at all Convenient | 0 | 1 | 1
  Missing | 5 | 3 | 8

4. Secondary Outcome: Subject Perceptions of Easypod: Preference to Use Easypod Over Two Other rhGH Pen Injection Devices.
Time Frame: 90 Days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Humatrope | Genotropin | Total
Number analyzed (Participants) | 16 | 19 | 35
Participants
  Strongly Agree | 2 | 6 | 8
  Agree | 2 | 2 | 4
  Neutral | 2 | 1 | 3
  Disagree | 2 | 3 | 5
  Strongly Disagree | 3 | 4 | 7
  Missing | 5 | 3 | 8

ADVERSE EVENTS:
Time Frame: Day 1, Week 12 and Four Week Follow-up
Arm/Group | Log Aware | Log Unaware
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 2/21 | 5/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Log Aware (N=21) | Log Unaware (N=21)
Brainstem Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncopal episodes (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Log Aware (N=21) | Log Unaware (N=21)
Constipation (Gastrointestinal disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Back Injury (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Enrollment ended early due to slow enrollment. Only 44 enrolled of the 100 subjects needed. Of the 44 enrolled, only 35 subjects had valid device data for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution or Principal Investigator can publish or present any results to a third party until (i) EMD Serono publishes the results (ii) Institution receives notification from EMD Serono that publication is no longer planned (iii) 18 months following the completion of the study whichever occurs first. Prior to publishing or presenting results, the Principal Investigator needs to provide EMD Serono with a copy of the presentation for review and approval.